CLINICAL TRIAL: NCT02988479
Title: Out-of Pocket Payments in Patients With Primary Lymphedema in France and Inequities of Access to Healthcare
Brief Title: Out-of Pocket Payments in Patients With Lymphedema
Acronym: Lymphorac2
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: 9638
Record Dates: First submitted 2016-09-02; First posted 2016-12-09 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Primary Lymphedema
MeSH Terms: conditions — Lymphedema | interventions — Health Expenditures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Out of pocket payments in patients

SUMMARY:
Primary lymphedema is a chronic condition posing a high burden on patients. Clinical guidelines emphasize the role of compression therapy by prescription medical devices. Even in a mandatory publicly funded health insurance system, out-of-pocket payments (OOPP) may exist due to the price and reimbursement setting processes. OOPP may threaten the equity of care and drive patients to forgo care. The investigators aim was to analyze the distributive effects of OOPP for primary lymphedema patients in France.

A prospective, multicenter study will be conducted in France in 2015 on patients with primary lymphedema. Household ability to pay will be specified by net income and OOPP will be assessed prospectively over 6 months for outpatient care (visits, drugs, medical devices, nursing care, biological tests, imaging, physiotherapy and transportations). Both mandatory and voluntary health insurance reimbursements will be considered. The investigators will combine concentration curves and concentration indices to assess the distributive effects.

ELIGIBILITY:
Inclusion criteria:

* Patient aged over six years, with primary lymphedema, regardless of the severity of the disease;
* Patient treated in one of the centres participating in the study;
* Patient (and her legal representative for minors) who gave her written consent [or did not refuse to participate, according to local Law];
* Patient with Internet access and an active email address.

Exclusion criteria:

* Patients with concomitant chronic venous insufficiency;
* Patient not covered by any health care insurance scheme;
* People protected under the law.

Ages: 6 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All consecutive patients meeting the inclusion criteria will be included in each participating centre during the inclusion phase
Sampling Method: Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
The mean monthly out-of-pocket payment as assessed by an online self-questionnaire | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Gregoire MERCIER, MD, PHD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- University Hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mercier G, Pastor J, Clement V, Rodts U, Moffat C, Quere I. Out-of-pocket payments, vertical equity and unmet medical needs in France: A national multicenter prospective study on lymphedema. PLoS One. 2019 May 8;14(5):e0216386. doi: 10.1371/journal.pone.0216386. eCollection 2019. PMID 31067244